CLINICAL TRIAL: NCT03550248
Title: Healthy Weights for Children Project (Phase 3)
Brief Title: Healthy Together Program Evaluation (Phase 3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government); The Bridge Youth and Family Services, Kelowna, BC, Canada (Unknown)
Responsible Party: Principal Investigator, Joan Bottorff, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1415-HQ-000616.
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Health Knowledge, Attitudes, Practice; Overweight and Obesity
Keywords: Healthy Weights; Health Promotion; Scale-up; Family Health; Prevention; Childhood Obesity; Physical Activity; Cooking Activity; Family education model
MeSH Terms: conditions — Behavior; Overweight; Obesity; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participating organizations will deliver the Healthy Together (HT) program to children/youth and their parents/caregivers. Participants in the program will be invited to complete questionnaires to evaluate the program at mid point (after 15 sessions) and post program (after 30 sessions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Other): Participants will receive the intervention - Healthy Together (HT).
  Interventions: Behavioral: Healthy Together

INTERVENTIONS:
Behavioral: Healthy Together — The Healthy Together (HT) program is designed to reduce overweight and obesity among children and youth in priority populations such as Indigenous, immigrant and refugee, and low income families.The HT program consists of 30 sessions, each of which includes cooking and eating together, physical activity and a learning activity covering topics that promote healthy weights. The HT program is delivered by trained facilitators who are provided with a program manual and resources. Trained facilitators in participating community organizations offer the HT program by integrating it within core programming.
  Other Names: Healthy Together Children's Health Program

SUMMARY:
Healthy Together is a program that promotes the achievement and maintenance of healthy weights in children and their families.

DETAILED DESCRIPTION:
The purpose of the Phase 3 scale up project is to expand the reach and impact of Healthy Together (HT), by supporting the integration of the HT program into core services of organizations serving children (up to 18 years) and families, particularly those from under-served populations across diverse communities and settings in Canada. The HT program offers a flexible, effective, integrated approach, relevant to multiple contexts, creating potential to become a sustainable approach to promoting healthier weights in Canadian children. The objectives of the evaluation for Phase 3 are to:

1. Describe the effectiveness of the HT program in relation to knowledge, attitude and behavior change at the individual, family, and community level.
2. Monitor quality and sustainability of HT, when offered as part of core service by organizations to meet diverse community needs and cultural contexts.
3. Create an effective knowledge mobilization framework to increase practice and policy influence of HT, in collaboration with regional, provincial and national networks.

ELIGIBILITY:
Community partner organizations with capacity and infrastructure to implement the HT program are eligible to be implementation sites. Priority is given to community organizations serving Indigenous, immigrants/refugees, low income/low literacy groups, and families residing in rural communities. All sites will be required to integrate HT into their existing services.

Inclusion criteria for each participant group are as follows:

Families: HT is designed for children (up to 18 years of age) and families. Children and families participating in programs offered by the partner organizations are eligible to attend HT. All interested families will be able to access the program regardless of their previous knowledge or skill level. Participants do not have to be overweight/obese to participate in sessions.

HT Facilitators: Staff members who are identified by the partner organizations, trained to implement the HT program and directly involved in HT program delivery will be eligible to participate in the evaluation.

Directors of Partner Organizations: Partner organizations will be asked to identify a director (supervisor) that has administrative responsibility for overseeing the delivery of services for children/families that includes the HT program.

National Advisory Committee (NAC): Members of the National Advisory Committee established by The Bridge Youth and Family Service Society for Phase 3 of this project.

Exclusion Criteria:

Family members who have not participated in any of the HT sessions offered as part of on-going services provided by the partner organization.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3400 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in Physical Activity Behaviour | At mid point in the HT program (i.e., following the first 15 weekly sessions) and at HT program completion (i.e., following the second set of 15 weekly sessions)
  Godin Physical Activity Leisure Time Questionnaire
Changes in Healthy Eating | At mid point in the HT program (i.e., following the first 15 weekly sessions) and at HT program completion (i.e., following the second set of 15 weekly sessions)
  Self-reported changes in eating behavior because of participation in the HT program using validated survey questions

SECONDARY OUTCOMES:
Knowledge of healthy diet and physical activity behaviors | At mid point in the HT program (i.e., following the first 15 weekly sessions) and at HT program completion (i.e., following the second set of 15 weekly sessions)
  Self-reported knowledge using validated survey questions

OTHER OUTCOMES:
Sustainability assessment (HT program implementation) | At HT program completion (i.e., following delivery of 30 weekly sessions) and 1 year follow-up
  Perceptions of HT program maintenance and sustainability from directors & facilitators - using semi-structured telephone interviews
Level of success in increasing practice and policy influence of the HT program | Year 1, 2, and 3
  Semi-structured interviews with Directors and National Advisory Committee Members

CONTACTS AND LOCATIONS:
Overall Officials: Joan L Bottorff, PhD, RN, Principal Investigator — University of British Columbia
Locations (1):
- Bridge Youth and Family Services, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bottorff JL, Huisken A, Hopkins M, Nesmith C. A RE-AIM evaluation of Healthy Together: a family-centred program to support children's healthy weights. BMC Public Health. 2020 Nov 23;20(1):1754. doi: 10.1186/s12889-020-09737-8. PMID 33225915